CLINICAL TRIAL: NCT00001205
Title: Natural History of Treated Neurocysticercosis and Long-Term Outcomes
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 850127; 85-I-0127
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-01-22 (Actual); Status verified 2026-01-16

CONDITIONS: Cysticercosis; Neurocysticercosis
Keywords: Tapeworm; Taenia Solium; Neurocysticercosis; Natural History; Seizures; Aseptic Meningitis; Hydrocephalus
MeSH Terms: conditions — Cysticercosis; Neurocysticercosis; Cestode Infections; Taeniasis; Seizures; Meningitis, Aseptic; Hydrocephalus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Arm 1: Subarachnoid (racemose) neurocysticercosis
- Arm 2: Ventricular without other viable disease
- Arm 3: Parenchymal cyst(s)--non-calcified parenchymal disease at time of referral
- Arm 4: Calcified parenchymal disease with symptoms (seizures)
- Arm 5: Calcified parenchymal disease without symptoms
- Arm 6: Endemic exposure--subjects with compatible epidemiologic exposure to T. solium

SUMMARY:
Neurocysticercosis is a brain disease due to the larval stage of the pork tapeworm (Taenia solium). The most common symptoms patient experience from infection inside the substance of the brain (parenchymal disease) are seizures and headaches. When the infection is either inside the fluid pockets inside the brain (ventricular disease) or in the space around the brain (subarachnoid disease) patients can have chronic headaches, relapsing aseptic meningitis, hydrocephalus, stroke, and may require neurosurgical intervention. The purpose of this study is to treat patients with anthelmintic therapy (praziquantel and/or albendazole) and anti-inflammatories in alignment with currently accepted best practices and guidelines, depending on the neurocysticercosis subtype. The purpose of the study is to better understand and characterize clinical, biologic, and management factors during treatment that influence long term outcomes. In order to understand this further we collect patient clinical information, patient survey responses, blood, urine samples, and additional cerebral spinal fluid if already being collected for clinical care....

DETAILED DESCRIPTION:
Study Description:

The purpose of this protocol is to follow participants with cysticercosis during and after completion of treatment, to characterize the disease course during both short- and long-term follow-up, assess biomarkers associated with infection and response to treatment, improve diagnostic assays, and explore host-parasite interactions.

Primary Objective:

The primary objective is to characterize the biochemical and clinical course of neurocysticercosis (NCC) during and after treatment with long-term follow-up.

Secondary Objectives:

1. To develop novel biomarkers associated with active infection
2. To further understand host-parasite interactions, including the inflammatory response
3. Understand the basis for the pleiomorphic clinical manifestations, including the possible contributions of parasite and host genetics
4. Develop a screening paradigm

Primary Endpoint:

Description of clinical presentation, imaging features, morbidity, response to treatment, and outcomes in all forms of NCC.

Secondary Endpoints:

1. Central and peripheral immune cell phenotyping and cytokine measurements
2. Including, but not limited to bulk transcriptomics, referral to study for participant whole genome sequencing, cestode-specific genome sequencing
3. Biobanking cerebrospinal fluid (CSF), serum, plasma, urine
4. Test known and novel biomarkers, serologic responses in the pre-clinical stage of neurocysticercosis, correlate findings with imaging.

ELIGIBILITY:
* INCLUSION CRITERIA:

Arms 1-5 (NCC):

1. Aged 3 years and older.
2. Ability of participant (or legally authorized representative, LAR) to understand and the willingness to sign a written informed consent document.
3. Patients with proven or likely NCC

Arm 6 (Endemic Exposures):

1. Patient with epidemiologic history compatible with possible exposure to NCC
2. Aged 18 years and older.

EXCLUSION CRITERIA:

Not applicable

Ages: 3 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1. Arms 1-5 (neurocysticercosis arms): male and female subjects over age 3 years with likely or definite neurocysticercosis (NCC) diagnosis 2. Arm 6 (endemic exposure arm): subjects 18 years or older with an epidemiologic history compatible with possible exposure to Taenia solium.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 1985-10-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to characterize the biochemical and clinical course of neurocysticercosis (NCC) during and after treatment with long-term follow-up. | Ongoing
  To study the clinical course of cysticercosis following therapy and diminish morbidity associated with treatment of cysticercosis including neurocysticercosis or the inflammation associated with therapy

SECONDARY OUTCOMES:
Central and peripheral immune cell phenotyping and cytokine measurements | 2-5 years
Test known and novel biomarkers, serologic responses in the pre-clinical stage of neurocysticercosis, correlate findings with imaging. | 2-5 years
Biobanking cerebrospinal fluid (CSF), serum, plasma, urine | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Elise M O'Connell, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] McAleese KR, Guzman JJ, Thumm L, Nutman TB, Showler A, O'Connell EM. Chagas Disease Prevalence in a Cohort of Neurocysticercosis Patients in a Nonendemic Setting. Clin Infect Dis. 2022 Sep 14;75(5):897-900. doi: 10.1093/cid/ciac076. PMID 35134144
- [Background] Beatty NL, Kaur H, Schlaffer K, Thompson K, Manavalan P, Rijos ZR, Raman AA, Droghini HR, O'Connell EM. Subarachnoid Neurocysticercosis Case Series Reveals a Significant Delay in Diagnosis-Requiring a High Index of Suspicion Among Those at Risk. Open Forum Infect Dis. 2024 Mar 21;11(5):ofae176. doi: 10.1093/ofid/ofae176. eCollection 2024 May. PMID 38680612
- [Background] Tang NL, Nash TE, Corda M, Nutman TB, O'Connell EM. Triplex ELISA for Assessing Durability of Taenia solium Seropositivity after Neurocysticercosis Cure. Emerg Infect Dis. 2023 Jul;29(7):1340-1348. doi: 10.3201/eid2907.230364. PMID 37347506
- [Background] Corda M, Sciurba J, Blaha J, Mahanty S, Paredes A, Garcia HH, Nash TE, Nutman TB, O'Connell EM. A recombinant monoclonal-based Taenia antigen assay that reflects disease activity in extra-parenchymal neurocysticercosis. PLoS Negl Trop Dis. 2022 May 26;16(5):e0010442. doi: 10.1371/journal.pntd.0010442. eCollection 2022 May. PMID 35617367
- [Background] Harrison S, Thumm L, Nash TE, Nutman TB, O'Connell EM. The Local Inflammatory Profile and Predictors of Treatment Success in Subarachnoid Neurocysticercosis. Clin Infect Dis. 2021 May 4;72(9):e326-e333. doi: 10.1093/cid/ciaa1128. PMID 33269789
- [Background] Nash TE, O'Connell EM. Subarachnoid neurocysticercosis: emerging concepts and treatment. Curr Opin Infect Dis. 2020 Oct;33(5):339-346. doi: 10.1097/QCO.0000000000000669. PMID 32868512
- [Background] Tang NL, Schaughency P, Gazzinelli-Guimaraes P, Lack J, Thumm L, Miltenberger E, Nash TE, Nutman TB, O'Connell EM. Immunologic Profiling of CSF in Subarachnoid Neurocysticercosis Reveals Specific Interleukin-10-Producing Cell Populations During Treatment. Neurol Neuroimmunol Neuroinflamm. 2024 Nov;11(6):e200320. doi: 10.1212/NXI.0000000000200320. Epub 2024 Oct 30. PMID 39475624
- [Background] Nash TE, O'Connell EM, Hammoud DA, Wetzler L, Ware JM, Mahanty S. Natural History of Treated Subarachnoid Neurocysticercosis. Am J Trop Med Hyg. 2020 Jan;102(1):78-89. doi: 10.4269/ajtmh.19-0436. PMID 31642423
- [Background] O'Connell EM, Harrison S, Dahlstrom E, Nash T, Nutman TB. A Novel, Highly Sensitive Quantitative Polymerase Chain Reaction Assay for the Diagnosis of Subarachnoid and Ventricular Neurocysticercosis and for Assessing Responses to Treatment. Clin Infect Dis. 2020 Apr 15;70(9):1875-1881. doi: 10.1093/cid/ciz541. PMID 31232448
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1985-I-0127.html